CLINICAL TRIAL: NCT01772602
Title: The National Amyotrophic Lateral Sclerosis Registry
Status: Recruiting | Type: Observational
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CDC-NCEH/ATSDR-5768
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Lou Gehrig's Disease; Motor Neuron Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this registry is to (A) better describe the incidence and prevalence of Amyotrophic Lateral Sclerosis (ALS) in the United States;(B) examine appropriate factors, such as environmental and occupational, that may be associated with the disease; (C) better outline key demographic factors (such as age, race or ethnicity, gender, and family history of individuals who are diagnosed with the disease) associated with the disease; and (D) better examine the connection between ALS and other motor neuron disorders that can be confused with ALS, misdiagnosed as ALS, and in some cases progress to ALS.

DETAILED DESCRIPTION:
The National ALS Registry's Research Notification System allows person with ALS to participate in clinical trials.

ELIGIBILITY:
Inclusion Criteria:

- U.S. citizens 18 years of age or older

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ALS cases in the United States
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2010-10; Primary Completion 2040-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
The National Amyotrophic Lateral Sclerosis (ALS) Registry | 1 year
  To determine the incidence and prevalence of Amyotrophic Lateral Sclerosis in the US.

SECONDARY OUTCOMES:
Risk factors of ALS | 1 year
  To learn more about the potential risk factors for ALS

CONTACTS AND LOCATIONS:
Overall Officials: Paul Mehta, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- CDC, Atlanta, Georgia, United States

REFERENCES:
- See also: Click here to enroll in the National ALS Registry — http://www.cdc.gov/als